CLINICAL TRIAL: NCT05822570
Title: Oxygen Dissociation Curve in Patients Undergoing Orthotopic Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: O2DO2 in LTX
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-11

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; Oxygen dissociation curve

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessment of Oxygen Dissociation Curve (ODC) — ODC will be assessed at 5 timepoints: T0 after installation of arterial catheter, T1 before clamping of the liver, T2 5-10 min before reperfusion of the liver graft, T3 45 min after reperfusion, T4 1 h after T3 or at end of surgery

SUMMARY:
Hemoglobin (Hb) is the molecule responsible for the transport of oxygen (O2) to the tissues in mammals.

The p50 and the Hill coefficient (HC) best describe the ODC. The interaction between Hb and O2 can be influenced by many agents and conditions like temperature, pH, pCO2 and 2,3-diphosphoglycerate (2,3-DPG).

During liver transplantation numerous profound physiological changes occur, linked to the different stages of the surgical procedure.

Previous studies in humans and animals undergoing liver transplantation have shown that while the ODC seems preserved during preparation and the anhepatic phase, a left shift of the ODC occurs after reperfusion . This left shift of the ODC could imply a decreased release of oxygen to the tissues, probably worsening hemodynamic instability.

With this pilot study the investigator aim to measure ODCs at baseline and at different stages during orthotopic liver transplantation in patients in order to get deeper understanding of oxygen delivery and supply during liver transplantation surgery.

DETAILED DESCRIPTION:
Hemoglobin (Hb) is the molecule responsible for the transport of oxygen (O2) to the tissues in mammals.

First described by Bohr at the beginning of the 20th century, the interaction between oxygen and hemoglobin is represented by the oxygen-hemoglobin dissociation curve (ODC), which has a sigmoid shape. The p50 and the Hill coefficient (HC) best describe the ODC. The p50 represents the partial pressure of O2 at which the 50% of Hb is saturated with O2, and the Hill coefficient represents the maximal steepness of the curve in the logarithmic Hill plot. The interaction between Hb and O2 can be influenced by many agents and conditions like temperature, pH, pCO2 and 2,3-diphospoglycerate (2,3-DPG)(1). An increase in p50 indicates a shift of the ODC to the right and a decrease in Hb-O2 affinity, whereas a decrease of the p50 indicates a shift of the ODC to the left and an increased affinity .

Liver disease, in particular liver cirrhosis, is thought to influence the ODC in many ways, a right shift due to a stimulation in the production of 2,3-DPG has been described. Also Caldwell et al. showed a right shift of the ODC for cirrhotic patients, although they couldn't demonstrate the reason for this shift and only postulated that the acid-base balance in the red blood cell or the cation concentration could be abnormal in these patients. Patients with End Stage Liver Disease (ESLD) show an hyperdynamic circulation, an adaptive reaction to a possible occult ischemia and splanchnic vasodilatation (8). Under physiological conditions, the oxygen consumption (VO2) is independent of oxygen delivery (DO2). When DO2 decreases under a critical level, oxygen extraction from hemoglobin can increase to maintain VO2. Under this critical DO2 level, as oxygen extraction has reached its maximum, VO2 will decrease, this state is called physiological oxygen supply dependency. It has been postulated that in some diseases and conditions, such as ARDS, sepsis, acute liver failure or extensive surgery, a pathological oxygen supply dependency may exist. When considering the whole oxygen supply, it has to be taken into account that measurements of DO2 and VO2 alone don't acknowledge the impact of the ODC on the effective delivery of oxygen in the tissue. Also under normal conditions where DO2 and VO2 are in the normal range, the oxygen extraction rate could be impaired by changes in the ODC. Orthotopic liver transplantation (OLT) is an important step in the therapy of end stage liver disease and represent a complex intervention, both from the surgical and anesthesiologic point of view. During liver transplantation numerous profound physiological changes occur, linked to the different stages of the surgical procedure. At first, in the preparation phase, the native liver and the vessels are dissected and bleeding may occur. In the second phase of OLT the inferior vena cava will be clamped, with resulting hemodynamic instability from reduced preload and congestion in the inferior part of the body. During this so called anhepatic phase lactate and other metabolisms end products accumulate. After anastomosis of the vena cava and the portal vein, the reperfusion phase begins. Here, due to the return in the circulation of acidotic blood and accumulated metabolites from the inferior part of the body, profound hemodynamic instability with decreased blood pressure can be observed. Previous studies in humans and animals undergoing liver transplantation have shown that while the ODC seems preserved during preparation and the anhepatic phase, a left shift of the ODC occurs after reperfusion . This left shift of the ODC could imply a decreased release of oxygen to the tissues, probably worsening hemodynamic instability.

With this pilot study the investigator aim to measure ODCs at baseline and at different stages during orthotopic liver transplantation in patients in order to get deeper understanding of oxygen delivery and supply during liver transplantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patien scheduled for LTX
* Age 18 years to 99 years
* Signed informed content form.

Exclusion Criteria:

* Known hemoglobinopathy
* Need for more than 3 packed erythrocytes before assessment at T4.
* preoperative predicted need for more than 3 based on study team
* MELD score < 10
* stay at high attitude (>3000 m) for more days over the last 4 weeks

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for orthotopic liver transplantation
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Oxygen Dissocation Curve | 24 hours
  Oxgen delivery curve characteristics based on p50 values, Hill-coefficient and 2,3 DPG

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided